CLINICAL TRIAL: NCT04450680
Title: A Prospective Cohort Study on Beta-lactam Therapeutic Drug Monitoring in Singapore
Brief Title: Beta-lactam Therapeutic Drug Monitoring in Singapore
Acronym: BLAST-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BLAST-2
Record Dates: First submitted 2020-06-12; First posted 2020-06-29 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Beta-lactam Therapeutic Drug Monitoring — Monitoring serum beta-lactam levels to individualise beta-lactam doses and ensure therapeutic target attainment

SUMMARY:
This is a prospective cohort study to evaluate clinical utility and feasibility of beta-lactam therapeutic drug monitoring in Singapore. The investigators hypothesise that conventional beta-lactam dosing regimens based on manufacturer's recommendations (derived from Phase I studies on healthy volunteers) will produce sub-optimal levels in at least half of the patients. Hence, beta-lactam therapeutic drug monitoring and dose individualisation will be required for optimal clinical outcomes. The investigators' secondary aims include correlating various therapeutic targets with clinical outcomes to identify a suitable therapeutic target for clinical use and to characterise beta-lactam pharmacokinetics in sub-group of patients with complex pharmacokinetics so that local empirical dosing regimens can be formulated.

DETAILED DESCRIPTION:
Despite widespread use, conventional beta-lactam dosing regimens, derived from healthy volunteers, are sub-optimal clinically as patients display variable pharmacokinetics. This problem is further confounded by rising antimicrobial resistance and the need for high dose beta-lactams, exceeding licensed recommendations. In order to optimise beta-lactam therapy, dose individualisation using therapeutic drug monitoring (TDM) has been suggested. However, experience with beta-lactam TDM is limited with varying practices worldwide. Therapeutic targets are also variable and have not been extensively validated. Hence, this study primarily aims to establish clinical feasibility and utility of beta-lactam TDM. The investigators hypothesise that conventional beta-lactam dosing will produce sub-optimal levels in at least half of the patients, justifying need for TDM and dose individualisation to improve clinical outcomes. The secondary aims include correlating various therapeutic targets with clinical outcomes to identify a suitable therapeutic target for clinical use and to characterise beta-lactam pharmacokinetics and recommend local empirical dosing regimens.

The investigators propose a prospective cohort study on adult patients (≥21 years) admitted to SGH. Four blood samples will be obtained over a dosing interval and assayed using liquid chromatography with tandem mass spectrometry. Levels and dose adjustment recommendations will be reported to physicians by infectious disease pharmacists.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (21 years and above)
* Admitted to Singapore General Hospital
* Receiving beta-lactam therapy for documented or suspected infection
* Indication for beta-lactam therapeutic drug monitoring: critically ill, altered pharmacokinetics (burns, obese, on extracorporeal therapy, dialysis), immunocompromised, resistant pathogens, deep-seated infections, suspected or at risk for adverse effects

Exclusion Criteria:

* Expected mortality within next 24 hours
* Pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the above-mentioned hospital and receiving beta-lactam therapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
proportion of patients achieving beta-lactam therapeutic targets | until end of beta-lactam therapy, an average of 2 weeks
  proportion of patients achieving beta-lactam therapeutic targets

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Chua, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huttner A, Harbarth S, Hope WW, Lipman J, Roberts JA. Therapeutic drug monitoring of the beta-lactam antibiotics: what is the evidence and which patients should we be using it for? J Antimicrob Chemother. 2015 Dec;70(12):3178-83. doi: 10.1093/jac/dkv201. Epub 2015 Jul 17. PMID 26188037
- [Background] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437
- [Background] Roberts JA, Ulldemolins M, Roberts MS, McWhinney B, Ungerer J, Paterson DL, Lipman J. Therapeutic drug monitoring of beta-lactams in critically ill patients: proof of concept. Int J Antimicrob Agents. 2010 Oct;36(4):332-9. doi: 10.1016/j.ijantimicag.2010.06.008. Epub 2010 Aug 3. PMID 20685085
- [Background] Heffernan AJ, Sime FB, Lipman J, Roberts JA. Individualising Therapy to Minimize Bacterial Multidrug Resistance. Drugs. 2018 Apr;78(6):621-641. doi: 10.1007/s40265-018-0891-9. PMID 29569104

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04450680/Prot_SAP_001.pdf